CLINICAL TRIAL: NCT00619190
Title: An Open Label Study of Aripiprazole in Children and Adolescents With Autism Spectrum Disorders
Brief Title: Study of Aripiprazole to Treat Children and Adolescents With Autism
Acronym: PAIRS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Linmarie Sikich, MD, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-1792 GCRC-2491
Record Dates: First submitted 2008-02-07; First posted 2008-02-20 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-02

CONDITIONS: Autistic Disorder; Asperger Syndrome; Autism Spectrum Disorder
Keywords: open label; aripiprazole; children; adolescents; autism spectrum disorders
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome; Autism Spectrum Disorder | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- open aripipraprazole (Experimental): Openly provided, flexibly dosed aripiprazole in doses from 1mg to 30mg
  Interventions: Drug: aripiprazole
- no medication control (No Intervention): group of children whose parents do not want them to take medications for autism over the year following enrollment in the trial.

INTERVENTIONS:
Drug: aripiprazole — aripiprazole, open label, flexibly dosed from 1mg to 30mg, provided for up to 12 months
  Other Names: Abilify
  Arms: open aripipraprazole

SUMMARY:
The purpose of this open label study in children and adolescents is to examine the acute and long-term effects of aripiprazole on problem behaviors associated with autism spectrum disorders and development in areas which appear to be affected by autism spectrum disorders.

DETAILED DESCRIPTION:
The purpose of this open label study in children and adolescents with autism spectrum disorders (ASD) is to examine the acute (12 week) and long-term (1 year) effects of aripiprazole on problem behaviors associated with ASD and development in three behavioral domains which appear particularly affected by ASD. We are also examining the safety and tolerability of aripiprazole in a range of children with autism. 20 children will be enrolled in the treatment part of the study. An additional 10 children, self selected by guardian desire not to pursue pharmacological treatment, will serve as a nonrandomized control group. This group will be provided with support but not any other treatments, come in for fewer visits and will be asked not to seek pharmacologic treatment outside the study. As of January 2010, we have completed enrollment in the treatment arm. Currently, we are only looking to enroll individuals in the control arm in which participants would not take any psychiatric medication.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between 30 months and 17 years 11 months, male or female, of any ethnicity and of any cognitive level
* Meet criteria for diagnosis of autism, Asperger's Disorder or Pervasive Developmental Order NOS (i.e. an autism spectrum disorder) based on clinical evaluation and either the Autism Diagnostic Interview - Revised (ADI-R) or the Autism Diagnostic Observation Scale (ADOS)
* Have a guardian who is able and willing to give written informed consent
* If competent, subject able and willing to give written assent for their own participation
* If on anticonvulsants, subject have been seizure-free and on a stable anticonvulsant regimen for at least 6 months
* Subjects may receive other nonpharmacologic treatment including dietary treatments

Exclusion Criteria:

* Diagnosis of Rett's syndrome or Child Disintegrative Disorder
* Taken psychotropic medications other than clonidine or diphenhydramine within 2 weeks
* Previous trial of aripiprazole
* Pregnant or nursing
* Epilepsy or another significant chronic medical illness

Ages: 30 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2006-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linmarie Sikich, MD, Principal Investigator — University of North Carolina, Department of Psychiatry
Locations (1):
- University of North Carolina, Department of Psychiatry, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open Aripipraprazole | no Medication Control
Started | 21 | 9
Completed | 20 | 9
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- no Medication Control: group of children whose parents do not want them to take medications for autism over the year following enrollment in the trial. They may receive behavioral interventions
- Total: Total of all reporting groups
Arm/Group | Open Aripipraprazole | no Medication Control | Total
Number analyzed (Participants) | 21 | 9 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 9 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.269 (3.75) | 11.11 (4.5) | 9.542 (4.272)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 19 | 8 | 27
Region of Enrollment [Number; unit: participants]
  United States | 21 | 9 | 30

OUTCOME MEASURES:

1. Secondary Outcome: Clinical Global Impressions Scale - Severity Score (CGI-S)
Description: One of the most widely used of clinician assessment tools in psychiatry, the CGI is an observer-rated scale that measures illness severity (CGI-S).
  The CGI is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (among the most severely ill patients).
Time Frame: Baseline to 12 weeks
Population: Only 20 out of 21 total participants was analyzed in the aripriprazole group because one participant dropped out before 12 weeks and so the data was not available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Aripipraprazole | no Medication Control
Number analyzed (Participants) | 20 | 9
units on a scale | 5.35 (0.74) | 4.5 (0.85)

2. Primary Outcome: Change From Baseline in Aberrant Behavior Checklist-Irritability at 12 Weeks
Description: The Aberrant Behavior Checklist (ABC) is a caregiver rated questionnaire for assessing problem behaviors of children over the past week relative to typically developing children of the same age. Problem behaviors are rated on a categorical scale between 0 not at all a problem and 3 problem is severe in degree. Raters are instructed to consider both the severity and the frequency of the behavior in determining how severe a problem the behavior is. Thus, if a given behavior occurs more often than in other children of the same age and sex, scores greater than or equal to 1 are warranted. The total score can range from a minimum of 0 (no problem behaviors) to a maximum of 174, higher the number the worse the symptoms.The irritability subscale consists of 15 items with a minimal score of 0 - no irritability problems to 45 - all irritability items rated as severe. A rating of 18 or more on the irritability subscale is considered clinically significant.
Time Frame: Baseline to 12 weeks
Population: Only 20 out of 21 total participants were analyzed in the aripriprazole group because one participant dropped out before 12 weeks and so the data was not available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Aripipraprazole | no Medication Control
Number analyzed (Participants) | 20 | 9
units on a scale | 7.6 (9.7) | -0.6 (0.50)

3. Secondary Outcome: Change From Baseline in the Aberrant Behavior Checklist -Lethargy/Social Withdrawal Subscale at 12 Weeks
Description: The Aberrant Behavior Checklist lethargy/social withdrawal subscale (ABC-SW) is the sum of ratings from 0 - not a problem at all to 3 - problem is severe in degree on 16 items within the Aberrant Behavior checklist (also described in the primary outcome measure section above). Scores can range from 0 to 48, with higher scores indicating more severe problems. The period for the rating is one week and the reference group is typically developing children of the same age and gender as the participant. Both frequency of the behaviors and severity of the problems related to them are considered. High ratings on these items reflect lack of response and interaction with other people in the child's environment.
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Aripipraprazole | no Medication Control
Number analyzed (Participants) | 20 | 9
units on a scale | -4.5 (6.4) | -0.3 (2.4)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from baseline to 12 weeks treatment. It was a systematic assessment of adverse effects.
Arm/Group | Open Aripipraprazole | no Medication Control
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/9
Other Adverse Events (participants affected / at risk) | 19/21 | 5/9
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Aripipraprazole (N=21) | no Medication Control (N=9)
Agitation (Psychiatric disorders) | 2 (21) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (21) | 1 (1)
Appetite Increased (Gastrointestinal disorders) | 4 (6) | 0 (0)
Appetite Decreased (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (General disorders) | 5 (7) | 1 (1)
Encopresis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Infection (Infections and infestations) | 7 (7) | 0 (0)
Fever (Infections and infestations) | 1 (1) | 2 (2)
Nightmares (General disorders) | 0 (0) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Headache/Migraine (General disorders) | 5 (5) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Allergies (Immune system disorders) | 0 (0) | 2 (2)
Mouth Sores (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No